CLINICAL TRIAL: NCT05498766
Title: Effect and Safety of Huaier Granule Versus SOX Regimen for the Prevention of Recurrence/Metastasis After Radical Surgery for Stage II-III Gastric Cancer Patients: a Prospective, Multi-center, Open-label and Randomised Control Study
Brief Title: Effect and Safety of Huaier Granule Versus SOX Regimen in Gastric Cancer Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, kaixiong tao, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE-202205
Record Dates: First submitted 2022-08-07; First posted 2022-08-12 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Gastric Cancer
Keywords: Huaier granule; Gastric cancer; SOX; Adjuvant therapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Tegafur; gimeracil; potassium oxonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huaier group (Experimental): The participants volunteering to take Huaier granule will be assigned to the Huaier group.
  Interventions: Drug: Huaier granule
- Control group (Active Comparator): The participants volunteering to take SOX will be assigned to the control group.
  Interventions: Drug: Oxaliplatin; Drug: Tegafur, Gimeracil and Oteracil Potassium

INTERVENTIONS:
Drug: Huaier granule — Huaier granule, oral administration, 10g each time, 3 times a day. Continuous medication until disease progression, the end of the study, intolerable toxicity, withdrawal from the study for any reason or death, or until the researcher determines that the participants will no longer benefit, whichever occurs first. After disease progression, whether to continue the medication or not should be determined by the researcher and participant together. Participants will start taking Huaier granule within 1 to 3 weeks after surgery.
  Other Names: Z20000109
  Arms: Huaier group
Drug: Oxaliplatin — Participants will receive intravenous infusion of 130 mg/m² oxaliplatin on the first day of treatment cycle.
  Arms: Control group
Drug: Tegafur, Gimeracil and Oteracil Potassium — Participants will receive oral Tegafur, Gimeracil and Oteracil Potassium (40 mg/m², twice a day) for 2 weeks, followed by 1 week of rest.
  Arms: Control group

SUMMARY:
This is a prospective, multi-center, open-label, randomised controlled study. The purpose of this study is to evaluate the efficacy and safety of Huaier Granule versus SOX regimen in the postoperative adjuvant treatment of resectable stage II-III gastric cancer.

DETAILED DESCRIPTION:
Gastric cancer (GC) is the second most frequently diagnosed cancer and the second leading cause of cancer related deaths in China. China has a higher mortality/incidence ratio (0.845). For stage II-III GC patients, the current standard treatment is D2 gastrectomy followed by adjuvant chemotherapy. Studies showed the 5-year survival rate of early GC is nearly 95%, while the 1-year recurrence and metastasis rate after surgery is about 50%, and the rate of 2-year is as high as 70%.

Although adjuvant chemotherapy can prevent recurrence, it is inevitable to the appearance of toxic and side effects, which seriously affect the prognosis and quality of life.

Traditional Chinese medicine plays a unique role in enhancement of immune function, detoxification, and synergism of chemoradiotherapy. Huaier granule is an extract from a medicinal fungus. Previous studies have shown that Huaier granule can inhibit the proliferation, angiogenesis, metastasis and invasion of cancer cells, and can reverse the resistance of targeted drugs. Previous studies demonstrated Huaier granule is benefit to resistance to recurrence and metastasis, prolongation of patients' survival, and improvement of quality of life.

In this study, about 30 research centers will participate. Total of 702 participants will be divided into two groups (the Huaier group and the control group) at a ratio of 1:1. The Huaier group will receive Huaier granule as postoperative adjuvant therapy, and the control group will receive SOX regimen. The planned length of patient recruitment enrolment will be 2 years and the total length of visits be 3 years. After enrollment, participants will be visited every 12 weeks (window period ± 14 days) until the end of the study or until the patient withdraws from the study for any reason or dies.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years
* Pathologically diagnosed as stage II or III gastric adenocarcinoma (including gastroesophageal junction).
* Receiving radical surgery (R0, D2 resection, more than 16 lymph nodes should be detected) for gastric adenocarcinoma within 2 months prior to enrollment, and not receiving adjuvant treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status from 0 to 2.
* Patients are volunteers, have signed informed consent, and agree to cooperate with investigators in data collection.

Exclusion Criteria:

* Patients had received neoadjuvant therapy.
* Patients who have received or plan to receive targeted therapy and/or immunotherapy。
* Patients allergic to the components of Huaier granules, or avoid to use Huaier granules or use with caution.
* More than two active primary tumors at the same time.
* Patients have not recovered from surgical complications after radical surgery.
* Patients received other Chinese patent medicine with anti-tumor effects.(including but not limited to Huaier Granule, Fufangbanmao Capsule, Huachansu Capsule, Kangai Injection, Pingxiao Table) in the past 1 month.
* Not able to take medication orally cause by difficulty in swallowing, complete or incomplete gastrointestinal obstruction, active bleeding from the gastrointestinal tract, perforation, etc.
* Pregnant or lactating women or women prepare for pregnancy.
* Serious concomitant infection disease.
* Patients with severe psychiatric illness or otherwise diseases are unsuitable for this study according to the judgment by investigators.
* Patients with combined immune disease and receiving immunosuppressive therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 702 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
3-year DFS rate | up to 36-months follow-up
  The proportion of patients who does not have recurrence of primary cancer, new gastric cancer, distant metastases (assessed by each investigator), or death from any cause within 3 years after receiving surgery.

SECONDARY OUTCOMES:
1, 2-year DFS rate | up to 12/24-months follow-up
  The proportion of patients who do not have recurrence of primary cancer, new gastric cancer, distant metastases (assessed by each investigator), or death from any cause within 1/2 years after receiving surgery.
1, 2, 3-year OS rate | up to 12/24/36-months follow-up
  The proportion of patients who will be alive within 1/2/3 years after receiving surgery.
1, 2, 3-year local recurrence-free survival rate | up to 12/24/36-months follow-up
  The proportion of patients who do not have local recurrence or regional lymph node metastasis from an cause within 1/2/3 years after receiving surgery.
1, 2, 3-year distant metastasis-free survival rate | up to 12/24/36-months follow-up
  The proportion of patients who do not have distant metastasis from an cause within 1/2/3 years after receiving surgery.
Quality of life score | Up to 36 months since the start of treatment
  The patients will evaluated by the Short-Form 36 (SF-36) Health Survey (Chinese version), which is a 36-item questionnaire measures health on 8 multi-item dimensions. Scores are computed for each dimension by adding the recorded item responses together and transforming the results onto a scale from 0 (worst health on scale) to 100 (best health on scale).
Incidence and severity of adverse events and serious adverse events | up to 36-months follow-up
  The incidence of adverse events and serious adverse events (referring to CTCAE 5.0 ) will be analyzed.
Incidence and severity of adverse reactions, serious adverse reactions, suspicious and unexpected serious adverse reactions | up to 36-months follow-up
  The incidence of ADR, SADR and SUSAR (referring to CTCAE 5.0 ) will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Kaixiong Tao, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (2):
- China (2):
  - Wuhan Union Hospital, Wuhan, Hubei
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong

IPD SHARING:
Plan to Share IPD: No